CLINICAL TRIAL: NCT02327195
Title: Active Emergence of From Isoflurane General Anesthesia Induced by Methylphenidate
Brief Title: General Anesthesia Emergence Induced by Methylphenidate
Acronym: MPOrtho
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nicoleta Stoicea (Other)
Responsible Party: Sponsor-Investigator, Nicoleta Stoicea, Research Scientist, Adj. Assistant professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013H0296
Record Dates: First submitted 2014-12-16; First posted 2014-12-30 (Estimated); Results first posted 2022-04-22 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Delayed Emergence From Anesthesia
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Experimental): Quillivant XR - Methylphenidate HCL Extended Release oral suspension - (after reconstruction with water - 5mg/mL) 20 mg (PO) given 2 hours prior to surgery
  Interventions: Drug: Methylphenidate HCl
- Placebo (Placebo Comparator): 20 mg Placebo (PO) given 2 hours prior to surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate HCl — Subjects will be randomly assigned to either the Methylphenidate or the Placebo arm, and be given a 20 mg dose (of Methylphenidate or Placebo) in liquid form (4 mL)
  Other Names: Concerta; Daytrana; Methylin; Ritalin
  Arms: Methylphenidate
Drug: Placebo — 20 mg of placebo (PO) will be given 2 hours prior to surgery
  Other Names: Placebo (PO)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether methylphenidate affects time of emergence from isoflurane general anesthesia. Time to emergence was defined as the time from termination of isoflurane to extubation. After stopping isoflurane infusion, when the patient breaths spontaneously with adequate tidal volume and respiratory rates, the trachea will be extubated and the time will be recorded.

DETAILED DESCRIPTION:
Based on this significant arousal stimulatory effect, the investigators hypothesize that methylphenidate (inhibitor of dopamine and norepinephrine transporters) decreases the emergence time from isoflurane general anesthesia.

PRIMARY OBJECTIVE:

To assess whether methylphenidate affects time of emergence from isoflurane general anesthesia. Time to emergence was defined as the time from termination of isoflurane to extubation. After stopping isoflurane infusion, when the patient breaths spontaneously with adequate tidal volume and respiratory rates, the trachea will be extubated and the time will be recorded.

SECONDARY OBJECTIVES:

* To assess the efficacy of methylphenidate in preventing post operative nausea and vomiting (PONV) by limited opioids consumption: PONV verbal response scale on a 0 to 10 verbally elicited scale: 0 (no nausea) to 10 (nausea as bad as it could be)
* To assess the efficacy of methylphenidate in preventing opioids dose escalation (fast cognitive improvement with efficient pain control -Postoperative Pain Numeric Rating Scale: O=None; (1-3)=Mild; (4-6)= Moderate; (7-10)=Severe).

Study Population: Adult patients at Ohio State University Wexner Medical Center - Sports Medicine, aged between 18-65 years, with an American Society of Anesthesiologists (ASA) physical status of I (normal healthy patient) or II (patients with mild systemic disease; no functional limitation) who are scheduled to undergo hip arthroscopic surgery - same day discharge - under isoflurane general anesthesia.

Single-center, prospective, randomized, double-blind, placebo-controlled trial involving 54 subjects scheduled to undergo arthroscopic orthopedic surgery under isoflurane general anesthesia at The Ohio State University Wexner Medical Center (OSUWMC) - University Hospital East. Eligible subjects that provide voluntary and written informed consent will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 65 years of age
* ASA I or II
* Capable and willing to consent
* Participants literate in English language

Exclusion Criteria:

* ADHD with current use of methylphenidate
* Hypersensitivity to methylphenidate
* ASA III, IV or V
* Patients with severe visual or auditory disorder
* Illiteracy
* Presence of a clinically diagnosed anxiety, agitation, major psychiatric condition such as bipolar disorder, uncontrolled major depression, schizophrenia
* Tics or Tourette's syndrome
* Glaucoma
* Hypertension, history of atrial arrhythmias (atrial fibrillation, atrial flutter), myocardial infarction
* Taking or have taken within the past 14 days a monoamine oxidase inhibitor or MAOI (Selegiline)
* Subjects who have participated or are currently participating in a clinical trial of an investigational drug within 30 days prior to surgery
* Any condition, which in the opinion of the investigator would make subject ineligible for participation in the study such as history of unstable cardiovascular, pulmonary, renal, hepatic, neurologic (seizures), hematologic or endocrine abnormality (hyperthyroidism, unstable Diabetes type I/II)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicoleta Stoicea, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methylphenidate | Placebo
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [25 to 40] | 36 [28 to 43] | 35 [28 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 10 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Emergence Time
Description: After stopping isoflurane infusion, when the patient breathes spontaneously with adequate tidal volume and respiratory rates, the trachea will be extubated and the time will be recorded.
Time Frame: From the moment when isoflurane infusion is stopped until time of extubation
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 27 | 27
minutes | 9 [5 to 13] | 9 [5 to 17]

2. Secondary Outcome: Number of Participants That Experienced Postoperative Nausea and Vomiting
Description: Efficacy of methylphenidate in preventing post operative nausea and vomiting (PONV) by limited opioids consumption: PONV verbal response scale on a 0 to 10 verbally elicited scale: 0 (no nausea) to 10 (nausea as bad as it could be)
Time Frame: First 24 Hours Postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 27 | 27
Participants | 5 | 3

3. Secondary Outcome: Opioid Dose Escalation Prevention
Description: Assess the efficacy of methylphenidate in preventing opioids dose escalation (fast cognitive improvement with efficient pain control -Postoperative Pain Numeric Rating Scale: O=None; (1-3)=Mild; (4-6)= Moderate; (7-10)=Severe).
Time Frame: During the length of hospital stay post surgery (on average 24 hours), and up to 3 days after surgery
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 27 | 27
Morphine Milligram Equivalents (MME) | 1.9 (4.6) | 2.8 (5.3)

ADVERSE EVENTS:
Time Frame: 34 days
Description: Continued multi-modal monitoring and vigilance with regard to any suspected adverse effects, including cardiovascular effects will help to fill the informational gap with regards to unknown cardiovascular side effects, emergence delirium incidence and perioperatory awareness.Due to the potential risk of drug related serious side effects, any clinical evidence of a serious adverse event will place the study on clinical hold until a full assessment and decision is made by the responsible parties.
Arm/Group | Methylphenidate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 11/27 | 11/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate (N=27) | Placebo (N=27)
Mild QTc prolongation (Cardiac disorders) | 11 (11) | 11 (11) — Mild QTc prolongation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT02327195/Prot_SAP_000.pdf